CLINICAL TRIAL: NCT03637413
Title: Effect of Hindmilk on Growth Velocity of Very Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Belal Alshaikh (Other)
Responsible Party: Sponsor-Investigator, Belal Alshaikh, Neonatologist, University of Calgary
Organization: University of Calgary (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB18-0195
Record Dates: First submitted 2018-08-14; First posted 2018-08-20 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Weight Gain
Keywords: preterm infants; hindmilk
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hindmilk (Experimental): Hindmilk, the milk at the end of a breast pumping session, has higher fat and energy content compared to the composite milk.
  Interventions: Dietary Supplement: Hindmilk

INTERVENTIONS:
Dietary Supplement: Hindmilk — Mother will be taught to separate her milk and infant will receive only hindmilk for feeds

SUMMARY:
Research question: Does feeding hindmilk improve weight gain in very preterm infants with poor growth velocity?

Hypothesis: In very preterm infants (born less than 32 weeks gestation) with poor postnatal growth velocity (<15 g/kg/day), feeding hindmilk would improve average weight gain by at least 4 g/kg per day.

Study design: This will be a prospective cohort study in very preterm infants admitted to the Neonatal Intensive Care Unit (NICU) at Foothills Medical Centre

DETAILED DESCRIPTION:
Extra-uterine growth restriction (EUGR) is one of the most common findings among very preterm infants at discharge from neonatal intensive care units. EUGR is associated with major morbidities such as bronchopulmonary dysplasia (BPD), retinopathy of prematurity (ROP) and impaired neurodevelopment. EUGR is caused by slow postnatal growth and largely results from energy and protein deficits. These deficits occur despite the current fortifications of human milk. Hindmilk, the milk at the end of a breast pumping session, has higher fat and energy content compared to the composite milk. Feeding hindmilk can be a natural and innovative way to provide additional calories for very preterm infant. Hindmilk is rich in some fatty acids that are currently under investigation to prevent BPD and ROP and improve neurodevelopment. The aim of this study is to assess growth benefits of feeding hindmilk and to explore whether it can improve fatty acids profile in very preterm infants.

Dietitians (RD) and Lactation Consultant (LC) will screen and identify eligible mother-infant pairs. Once mother's consent obtained, LC will hand out the "hindmilk information sheet" and teach the mother how to separate her milk. A sample (10 ml) of composite pumped fresh milk will be collected and placed in the fridge. These samples will be sent for analysis within 24 hours of collection to minimize any changes to contents. Samples for Erythrocyte membrane fatty acid (FA) profile will be collected on dried blood spot (30-100 µL). These samples will be collected within 72 hours of the consent. It will be coordinated with blood tests ordered by the clinical team within that period. Dried blood spots are stable in room temperature for 28 days however we will store them in the -80̊ C freezer within 72 hours of collection. Another milk sample, hindmilk this time, will be sent for testing within 24-48 hour of starting hindmilk. This is to ensure that assessment of milk contents is performed in the same mother's lactation stage. The second dried blood spot will be drawn after 2-4 weeks of starting hindmilk. The 2-4 weeks period is to allow timing with other blood work-ups. In General, blood glucose is done every 2-3 days in babies with poor growth and growth laboratory testing is normally done every 2-3 weeks.

Data on fluid volumes, feeds, macronutrients intakes and any change in nutrition plan will be collected from electronic dietitian's notes. Dietitians will ensure proper and detailed documentation of nutritional information. Average weight gain (in gram/kg per day) is calculated as mentioned before. Average weight gain will be compared initially between the week before and the week after starting hindmilk. The day that hindmilk started will be used to identify the start point however it will not be used in either the pre- or the post-hindmilk calculation. Clinical team will be encouraged to not order other changes to the nutrition plan for the first week after starting hindmilk. Daily weight, weekly length and head circumference will be collected from the electronic charts. Furthermore, weight, length and head circumference at completed gestational week will be used to calculate Z scores using Fenton Z scores calculator.

Data on maternal and neonatal characteristics will be collected from their electronic and physical charts. Composite milk, foremilk and hindmilk volumes will be collected from the collection sheet that has been already used in our NICU.

ELIGIBILITY:
Inclusion Criteria:

* Very preterm infant ( <32 weeks at birth)
* On full enteral feeds for more than 2 weeks (full feed is defined at the time of reaching 120 ml/kg/day with no parenteral nutrition used)
* Poor weight gain (<15 g/kg per day) despite optimization of energy and protein intakes by RDs (calories intake: 125-135 Kcal/kg per day and protein: 4-4.5 g/kg per day)
* Mothers have enough milk supply (>150% of infant's daily needs)

Exclusion Criteria

* Congenital anomalies
* Small for gestational age infants (< 10th percentile) at birth

Min Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-01-22 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Average Weight Gain | 2 weeks
  Difference in weight gain the week before hindmilk and the week after

SECONDARY OUTCOMES:
Effect of feeding hindmilk on anthropometrics | At 36 weeks post menstrual age and/or discharge (up to 13 weeks)
  Compared to published rates in NICUs
Effect of feeding hindmilk on body mass index | At 36 weeks post menstrual age and/or discharge (up to 13 weeks)
  Compared to published rates in NICUs
Incidence of extra uterine growth restriction | At 36 weeks post menstrual age and/or discharge (up to 13 weeks)
  Defined as wight less than 10th percentile. Compared to published rates in NICUs
Incidence of bronchopulmonary dysplasia and retinopathy of prematurity | At 36 weeks post menstrual age and/or discharge (up to 13 weeks)
  BPD will be defined according to Child Health and Human Development as the requirement for positive pressure support (CPAP or high flow nasal cannula ≥ 1 liter per minute (LPM)), or oxygen dependency at 36 corrected gestational age. ROP will be defined according to the international classification1 or requiring treatment. Compared to published rates in NICUs
Correlation between human milk content (fat, protein and energy) and weight gain | Within 4 weeks of enrollment
  Linear regression analysis will be used to correct for any confounding factors
Effect of hindmilk on erythrocyte membranes fatty acids profile. | Within 4 weeks of enrollment
  Comparison between sample taken at 24 hours and sample at week 2-4 after hindmilk
Changes in mother's milk volumes after feeding hindmilk. | Until 36 weeks post menstrual age and/or discharge (up to 13 weeks)
  Monitor the milk output of mothers throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Belal Alshaikh, MD, MSc, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT03637413/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT03637413/ICF_001.pdf